CLINICAL TRIAL: NCT03496571
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamic Effect of AK002 in Patients With Eosinophilic Gastritis and/or Eosinophilic Gastroenteritis
Brief Title: A Study of AK002 in Patients With Eosinophilic Gastritis and/or Eosinophilic Gastroenteritis
Acronym: ENIGMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-003
Record Dates: First submitted 2018-04-06; First posted 2018-04-12 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Gastroenteritis
Keywords: Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophil; EG; EGE; Eosinophilic gastrointestinal disorders; EGID
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects in this arm will receive 4 monthly doses of placebo.
  Interventions: Other: Placebo
- 1 mg/kg of AK002 (Experimental): Subjects in this arm will receive 4 monthly doses of AK002: a first dose of 0.3 mg/kg, a second dose of 1 mg/kg, a third dose of 1 mg/kg, and a fourth dose of 1 mg/kg
  Interventions: Drug: AK002
- 3 mg/kg of AK002 (Experimental): Subjects in this arm will receive 4 monthly doses of AK002: a first dose of 0.3 mg/kg, a second dose of 1 mg/kg, a third dose of 3 mg/kg, and a fourth dose of 3 mg/kg
  Interventions: Drug: AK002

INTERVENTIONS:
Drug: AK002 — AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8, a member of the CD33-related family of sialic acid-binding, immunoglobulin-like lectins (Siglecs).
  Arms: 1 mg/kg of AK002; 3 mg/kg of AK002
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, double-blind, randomized, placebo-controlled study to assess the effects of AK002, given monthly for 4 doses. It is hypothesized that AK002 is more effective than placebo control (alternative hypothesis) in reducing the number of eosinophils per high power field (HPF) in gastric and/or duodenal biopsies before and after receiving AK002 or placebo versus no difference between AK002 and placebo control (null hypothesis).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤80 years at the time of signing ICF.
2. Average weekly score of ≥3 (on a scale from 0-10, recorded for either abdominal pain, diarrhea and/or nausea on the PRO questionnaire during at least 2 out of 3 weeks of PRO collection. A minimum of four questionnaires must be completed each qualifying week.
3. Eosinophilia of the gastric mucosa ≥30 eosinophils/HPF in 5 HPFs and/or eosinophilia of the duodenal mucosa ≥30 eosinophils/HPF in 3 HPFs from the EGD performed during the screening period, without any other cause for the gastric eosinophilia (e.g., parasitic or other infection or malignancy).
4. Subjects must have failed or not be adequately controlled on standard-of-care treatments for EG or EGE symptoms (which could include PPIs, systemic or topical corticosteroids, and/or diet, among others).
5. If on other treatments for EG, EGE, or EoE at enrollment, stable dose for at least 5 half-lives prior to screening and willingness to continue on that dose for the duration of the study.
6. If subject is on pre-existing dietary restrictions, willingness to maintain dietary restrictions throughout the study, as much as possible.
7. Able and willing to comply with all study procedures.
8. Female subjects must be either post-menopausal for at least 1 year with FSH level >40 mIU/mL at screening or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer. Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant at any time during study participation.

Exclusion Criteria:

1. Known hypersensitivity to any constituent of the study drug.
2. Diagnosis of celiac disease or H. pylori infection as determined by screening EGD or a history of celiac disease diagnosed by prior EGD.
3. Presence of abnormal laboratory values considered by the Investigator to be clinically significant.
4. Grade 2 or higher lymphopenia (<0.8 × 109/L lymphocytes).
5. Any disease or condition (medical or surgical) or cardiac abnormality, which, in the opinion of the Investigator, would place the subject at increased risk.
6. History of malignancy; except carcinoma in situ in the cervix, early stage prostate cancer, or non-melanoma skin cancers. However, cancers that have been in remission for more than 5 years and are considered cured, can be enrolled (with the exception of breast cancer). All history of malignancy (including diagnosis, dates, and compliance with cancer screening recommendations) must be documented and certified by the Investigator, along with the statement that in their clinical judgment the tissue eosinophilia is attributable to EGID, rather than recurrence of malignancy.
7. Treatment with chemotherapy or radiotherapy in the preceding 6 months.
8. Treatment for a clinically significant helminthic parasitic infection within 6 months of screening and/or a positive helminthic test at screening.
9. Use of any medications that may interfere with the study such as immunosuppressive or immunomodulatory drugs (including azathioprine, 6-mercaptopurine, methotrexate, cyclosporine, tacrolimus, anti-TNF, anti-IL-5, anti-IL-5 receptor, dupilumab, anti-IgE antibodies, omalizumab) or systemic corticosteroids with a daily dose >10 mg of prednisone or equivalent, during 5 half-lives prior to screening or during the screening period, except for omalizumab taken in asthma and/or urticaria patients where their asthma and/or urticaria cannot be controlled on other medications. In such cases, the dose of omalizumab should remain stable during screening and throughout the study.
10. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives of the study drug administration.
11. Known history of alcohol, drug, or other substance abuse or dependence.
12. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to administration of study drug (or 90 days or 5 half-lives, whichever is longer, for biologic products).
13. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
14. Any other reason that in the opinion of the Investigator or Medical Monitor makes the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Director — Allakos Inc.
Locations (21):
- United States (21):
  - Phoenician Centers for Research and Innovation, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Ventura Clinical Trials, Ventura, California
  - UC Denver, Aurora, Colorado
  - Riverside Clinical Research, Edgewater, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Northwestern, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - National Institutes of Health, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Care Access Research, Pottsville, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Avant Research Associates, Austin, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dellon ES, Gonsalves N, Rothenberg ME, Hirano I, Chehade M, Peterson KA, Falk GW, Murray JA, Gehman LT, Chang AT, Singh B, Rasmussen HS, Genta RM. Determination of Biopsy Yield That Optimally Detects Eosinophilic Gastritis and/or Duodenitis in a Randomized Trial of Lirentelimab. Clin Gastroenterol Hepatol. 2022 Mar;20(3):535-545.e15. doi: 10.1016/j.cgh.2021.05.053. Epub 2021 Jun 2. PMID 34089846
- [Derived] Dellon ES, Peterson KA, Murray JA, Falk GW, Gonsalves N, Chehade M, Genta RM, Leung J, Khoury P, Klion AD, Hazan S, Vaezi M, Bledsoe AC, Durrani SR, Wang C, Shaw C, Chang AT, Singh B, Kamboj AP, Rasmussen HS, Rothenberg ME, Hirano I. Anti-Siglec-8 Antibody for Eosinophilic Gastritis and Duodenitis. N Engl J Med. 2020 Oct 22;383(17):1624-1634. doi: 10.1056/NEJMoa2012047. PMID 33085861

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Placebo
Started | 22 | 21 | 22
Completed | 20 | 19 | 20
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 22 | 65
Age, Continuous [Median (Full Range); unit: Years] | 39 [18 to 74] | 41 [20 to 67] | 36 [18 to 67] | 40 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 10 | 40
  Male | 5 | 8 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 5
  Not Hispanic or Latino | 21 | 17 | 22 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 21 | 17 | 22 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 21 | 22 | 65
Baseline Gastrointestinal Eosinophil Count [Mean (Standard Deviation); unit: Eosinophils/HPF] — Number of eosinophils per high power field (HPF) in gastric or duodenal mucosa
  Eosinophils/HPF | 101 (66) | 76 (40) | 74 (46) | 84 (52)
PRO Total Symptom Score (TSS) [Mean (Standard Deviation); unit: Score on a scale] — The PRO Total Symptom Score (TSS) is a patient-reported outcome (PRO) questionnaire comprises the following 8 symptoms: abdominal pain, nausea, vomiting, early satiety, loss of appetite, abdominal cramping, bloating, and diarrhea. Individual symptom scores ranged from 0 to 10. The daily total symptom score ranged from 0 to 80, with higher scores indicating greater severity. TSS score at the End of Study is the average of the daily scores from Days 85-99.
  Score on a scale | 34 (13) | 33 (14) | 29 (14) | 32 (14)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Number of Eosinophils Per High Power Field in Gastric or Duodenal Mucosa From Baseline
Description: Tissue eosinophil count obtained in biopsy specimens from the stomach and/or duodenum using esophago-gastro- duodenoscopy (EGD)
Time Frame: Baseline to Day 99
Population: Intention-to-treat
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Groups:
- Combined AK002: Combined group of 1 mg/kg of AK002 and 3 mg/kg of AK002.
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Combined AK002 | Placebo
Number analyzed (Participants) | 22 | 21 | 43 | 22
Percentage of Change | -79 [-95 to -59] | -92 [-100 to -81] | -86 [-94 to -71] | 9 [-15 to 31]
Statistical Analysis 1: Comparison: 1 mg/kg of AK002 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LSM Difference from Placebo = -95, 95% CI 2-sided [-122 to -68]
Statistical Analysis 2: Comparison: 3 mg/kg of AK002 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LSM Difference from Placebo = -102, 95% CI 2-sided [-128 to -76]
Statistical Analysis 3: Comparison: Combined AK002 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LSM Difference from Placebo = -98, 95% CI 2-sided [-121 to -76]

2. Secondary Outcome: Number of Treatment Responders
Description: Treatment Responders defined by >30% improvement in TSS and a reduction of >75% in eosinophils in gastric and/or duodenal mucosa. The eosinophil count is obtained on Day 99 and the TSS score is the average of the daily scores from Days 85-99.
Time Frame: On Days 85-99 and Day 99, respectively
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Combined AK002 | Placebo
Number analyzed (Participants) | 22 | 21 | 43 | 22
Participants | 13 | 14 | 27 | 1
Statistical Analysis 1: Comparison: 1 mg/kg of AK002 vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Percent Difference from Placebo = 55, 95% CI 2-sided [27 to 76]
Statistical Analysis 2: Comparison: 3 mg/kg of AK002 vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Percent Difference from Placebo = 62, 95% CI 2-sided [34 to 82]
Statistical Analysis 3: Comparison: Combined AK002 vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Percent Difference from Placebo = 58, 95% CI 2-sided [36 to 74]

3. Secondary Outcome: Percent Change in PRO Total Symptom Score (TSS) From Baseline
Description: The PRO Total Symptom Score (TSS) is a patient-reported outcome (PRO) questionnaire comprises the following 8 symptoms: abdominal pain, nausea, vomiting, early satiety, loss of appetite, abdominal cramping, bloating, and diarrhea. Individual symptom scores ranged from 0 to 10. The daily total symptom score ranged from 0 to 80, with higher scores indicating greater severity. TSS score at the End of Study is the average of the daily scores from Days 85-99.
Time Frame: Baseline to Days 85-99
Population: Intention-to-treat
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Combined AK002 | Placebo
Number analyzed (Participants) | 22 | 21 | 43 | 22
Percentage of Change | -42 [-56 to -28] | -55 [-70 to -40] | -48 [-58 to -39] | -22 [-37 to -7]
Statistical Analysis 1: Comparison: 1 mg/kg of AK002 vs Placebo; Test type: Superiority; p = 0.05, ANCOVA; LSM Difference from Placebo = -20, 95% CI 2-sided [-40 to 0]
Statistical Analysis 2: Comparison: 3 mg/kg of AK002 vs Placebo; Test type: Superiority; p = 0.002, ANCOVA; LSM Difference from Placebo = -33, 95% CI 2-sided [-53 to -13]
Statistical Analysis 3: Comparison: Combined AK002 vs Placebo; Test type: Superiority; p = 0.004, ANCOVA; LSM Difference from Placebo = -26, 95% CI 2-sided [-44 to -9]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 113
Arm/Group | 1 mg/kg of AK002 | 3 mg/kg of AK002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22 | 2/21 | 3/22
Other Adverse Events (participants affected / at risk) | 20/22 | 15/21 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/kg of AK002 (N=22) | 3 mg/kg of AK002 (N=21) | Placebo (N=22)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mental Status Change (Psychiatric disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron def anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/kg of AK002 (N=22) | 3 mg/kg of AK002 (N=21) | Placebo (N=22)
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 10 | 5
Headache (Nervous system disorders) | 3 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Fatigue (General disorders) | 3 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 2
White blood cell count increased (Investigations) | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT03496571/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03496571/SAP_001.pdf